CLINICAL TRIAL: NCT05425160
Title: Effects of Chair Rise and Step Ups on Cardiopulmonary Parameters Among Preserved Ejection Heart Failure Patients
Brief Title: Chair Rise and Step Ups on Cardiopulmonary Parameters Among Preserved Ejection Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iqra Arbab
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive lower limb activities (Chair rise and Step ups) (Experimental): Chair rise and Step ups Exercises
  Interventions: Other: Progressive lower limb activities (Chair rise and Step ups)
- Standard aerobic exercise i.e. low intensity walking (Active Comparator): aerobic exercise i.e. low intensity walking
  Interventions: Other: Standard aerobic exercise i.e. low intensity walking

INTERVENTIONS:
Other: Progressive lower limb activities (Chair rise and Step ups) — Progressive lower limb activities (Chair rise and Step ups) were be carried out weekly for upto 6 weeks. Before initiation, cardiopulmonary parameters i.e. Heart rate, oxygen saturation, cardiac output and stroke volume were measured at baseline and later at the termination of activity on each week. Initially, five repeated chair rise were conducted through SPPB and the time was noted to complete the task and step ups through 6MWD for a total period of 30 min. Lastly, fatigue component was assessed via FAS.
  Arms: Progressive lower limb activities (Chair rise and Step ups)
Other: Standard aerobic exercise i.e. low intensity walking — Standard aerobic exercise i.e. low intensity walking were conducted in both the groups. Follow up phone calls and 1 OPD visit were scheduled accordingly
  Arms: Standard aerobic exercise i.e. low intensity walking

SUMMARY:
To determine the effects of Chair Rise and Step ups on cardiopulmonary parameters among Preserved ejection Heart Failure Patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Preserved ejection Heart Failure Patients
* Both male and female
* Age > 60 years
* Preserved ejection fraction ≥ 45 %
* HF Duration ≥4 years

Exclusion Criteria:

* End stage heart failure
* Acute coronary syndrome
* Functional status limited due to condition other than heart failure
* Inability to adhere to study protocols.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | 6th week
  Changes from the baseline ; It is a 21 item paper self administered questionnaire. It aims to measure the extent to which HF prevents patients from living the way they would want to. The MLHFQ has been the most widely used instrument for evaluating HRQL in HF patients internationally. Five years ago, the MLHFQ was identified as the questionnaire with the best properties and even now it has the highest scores for reliability, and a good ability to both measure its objective (validity) and detect change over time
Short Physical Performance Battery (SPPB) | 6th week
  Changes from the baseline ; The SPPB is composed of 3 components-standing balance, gait, speed, and timed repeated chair rise-each scored on a scale from 0 to 4 and combined for a total score of 0 to 12. This protocol consisted of 3 types of progressive activities. Each type contains 2 to 4 tasks, performed in a single attempt. The protocol was performed in 30-minute sessions once a week. It was used to conduct chair rise activity only. Participant was asked to complete five chair stands and the time was noted and scored from 0-4 respectively.
6 Min Walk Distance (6MWT) | 6th Week
  Changes from the baseline ; The 6 min walk test (6MWT) is a functional performance measure to examine the functional status of patients with heart and lung disease. This protocol has 1 item only. It was completed in less than 10 minutes. A 6MWT distance of 300 m was also recently found to be a significant predictor of all-cause mortality in a multivariate model examining predictors of clinical outcome in elderly patients with advanced HF. Patients were instructed to cover the greatest distance possible during the allotted time, at a self-determined walking speed, and were allowed to pause and rest when needed. The distance covered was measured by a body-borne pedometer with which the total number of steps taken during the 6MWT were used to calculate the 6MWT distance using the equation reported by Roul et al. (d ¼ y × 10 m/x; where d ¼ distance ambulated in m; y ¼ total number of steps during 6MWT; and x ¼ number of steps for each subject to cover 10 m
Fatigue Assessment Scale (FAS) | 6th Week
  Changes from the baseline ; The FAS is a 10-item scale evaluating symptoms of chronic fatigue. The FAS is a self-report, paperand-pencil measure requiring approximately 2 min for administration. The scale has been validated in a population of both male and female. Each item of the FAS is answered using a five-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse-scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
Heart Rate | 6th week
  Changes from the baseline ; Heart rate was measured per minute through cardiac monitor
Oxygen Saturation | 6th week
  Changes from the baseline ; The saturation of arterial blood with oxygen as measured by pulse oximetry, expressed as percentage.
VO2 Max | 6th week
  Changes from the baseline ;The maximum or optimum rate at which the heart, lungs and muscles can effectively use oxygen during exercise, used as a way of measuring a person's individual aerobic capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Armed Forces Institute of Cardiology AFIC, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No